CLINICAL TRIAL: NCT05497232
Title: Clinical Analysis of Simultaneous Pancreas-kidney Transplantation for End-stage Renal Disease Associated With Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-hg-ks-17
Record Dates: First submitted 2022-08-06; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus；Uremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the homolateral simultaneous pancreas and kidney transplantation (Experimental): SPK using the surgical technique was performed in our department from September 2016 to January 2023 in the Department of Transplantation of the Second Affiliated Hospital of Guangzhou Medical University.
  Interventions: Procedure: simultaneous pancreas-kidney transplantation

INTERVENTIONS:
Procedure: simultaneous pancreas-kidney transplantation — Renal transplants were performed to the right external iliac artery and vein, and the ureter was anastomosed to the recipient ureter by using end-to-end anastomoses techniques. All the renal allografts were placed into retroperitoneum.
  Enteric drainage of exocrine secretions was performed on all pancreas transplants, systemic venous outflow (postcava), and arterial reconstruction with "y" graft (iliac artery). Lastly in all cases of renal transplant, the artery was anastomosed in all cases. The pancreas was placed intra-abdominally in all cases.

SUMMARY:
The first pancreas transplantation was performed in 1966, by 2015, more than 40,000 pancreas transplantation have been performed worldwide. Nevertheless, only several Chinese organ transplant centers carry out SPK because of surgery complications. simultaneous pancreas-kidney transplantation is a new and promising therapeutic option for the treatment for type 1 diabetes mellitus patients and end-stage renal disease. the preliminary treatment results are summarized to promote the further development of this work in China.

DETAILED DESCRIPTION:
simultaneous pancreas-kidney transplantation using the surgical technique was performed in our department from September 2016 to January 2023 in the Department of Transplantation of the Second Affiliated Hospital of Guangzhou Medical University. Patients were followed up for 2 to 36 months to summarize the efficacy and complications. we examined the influence of SPK on patient and graft survivals.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Diabetes patients with end-stage renal disease;
2. First time receiving SPKT;

Exclusion Criteria:

1. Pulmonary infection, urinary tract infection, hematuria CMV or BK virus infection occurred during treatment;
2. Using a large number of abnormal biological products (blood transfusion, plasma or coagulation factors) may contain foreign DNA;
3. Loss of graft due to thrombosis or AR;
4. Patients who are pregnant or have malignant tumors or patients with a history of cell therapy, whose tumor signals interfere with dd-cfDNA detection;
5. Patients who have poor compliance during treatment or suffer from mental illness.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient survival & pancreas graft survival & renal graft survival | 12 months
  Renal graft survival was defined as the exclusion of graft resection, restoration of dialysis, and death with graft function. Survival of the transplanted pancreas excluded resection of the transplanted pancreas, recovery of preoperative insulin dosage and death with graft function.

CONTACTS AND LOCATIONS:
Locations (1):
- 1Department of Organ Transplantation, Second Affiliated Hospital of Guangzhou Medical University,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
yes